CLINICAL TRIAL: NCT02587052
Title: A 1-year Comparison of Generic Tacrolimus (Tacni) and Prograf in Renal Transplant Patients - a Retrospective Matched Pair Analysis
Brief Title: A 1-year Comparison of Generic Tacrolimus (Tacni) and Prograf in Renal Transplant Patients - a Retrospective Matched Pair Analysis, GenTac
Acronym: GenTac
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015-08-01
Record Dates: First submitted 2015-10-19; First posted 2015-10-27 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2020-12

CONDITIONS: Renal Transplantation
Keywords: biopsy-proven acute rejection; graft loss; graft survival
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tacrolimus: 100 patients treated with generic tacrolimus
  Interventions: Drug: Generic tacrolimus
- Prograf: 100 patients treated with Prograf
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Generic tacrolimus — Generic tacrolimus
  Groups: Tacrolimus
Drug: Prograf — Prograf, the original tacrolimus
  Groups: Prograf

SUMMARY:
This is a retrospective analysis of two different cohorts of patients that has undergone renal transplantation. This is a matched pair analysis of 100 patients treated with generic tacrolimus that will be compared with 100 matched controls treated with Prograf. Data will be obtained from patients' charts, from the Swedish National Kidney Registry and from a local registry at Transplantationscentrum. Patients included in the study are patients receiving a first single kidney transplant from a deceased or a living donor, treated with Prograf or Tacni and transplanted between transplanted January 2012 and August 2014. The 1-year-outcome of patients following renal transplantation, including BPAR, serious adverse effects and graft survival will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a first single kidney transplant from a deceased or a living donor.
* Patients treated with Prograf or or generic tacrolimus
* Patients transplanted between 1 October 2012 and 1 August 2014

Exclusion Criteria:

* Multi-organ transplants
* Re-transplantations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is a retrospective analysis of two different cohorts of patients that have undergone renal transplantation at Transplanationscentrum in Gothenburg, Sweden. Approximately 100 patients treated with generic tacrolimus will be compared with 100 matched controls. The controls will be selected among 200 patients that are treated with Prograf. The matching will be based upon living/deceased, age of the donor, age of the patient and number of previous transplantations.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Biopsy-proven acute rejection (BPAR) | 1 year
Graft loss | 1 year
Death | 1 year

SECONDARY OUTCOMES:
Compare the following parameters in the two groups • Graft survival at 6 and 12 months • BPAR at 6 and 12 months • Calculated GFR at 12 months | 6 months, and 1 year
Compare serious adverse events at 12 months in the two groups | 1 year
Compare the the cost of admissions for rejection treatment in the two groups | 1 year
Tacrolimus dose at day of discharge | day of discharge, approx 7 days
Tacrolimus levels at day of discharge | day of discharge, approx 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Per Lindnér, MD, Principal Investigator — Transplant Center, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Transplant Institute, Sahlgrenska University Hospital, Gothenburg, Sweden